CLINICAL TRIAL: NCT07208851
Title: Development, Feasibility, and Acceptability of a One-time Problem Management Plus (PM+) Booster Session in the Bahamas: A Pilot Randomized Controlled Trial
Brief Title: Developing a Booster Session for Problem Management Plus in the Bahamas: A Pilot Randomized Controlled Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The New School (Other)
Responsible Party: Principal Investigator, Caroline McEneaney, PhD Candidate, Clinical Psychology, The New School
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-352-1244
Record Dates: First submitted 2025-09-27; First posted 2025-10-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-09

CONDITIONS: Depression Symptoms; Anxiety Symptoms
Keywords: PM+; Task-sharing interventions; Scalable mental health; Global mental health; Bahamian Mental Health; Hurricane; Climate Change
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Each participant will receive the full PM+ program (5 individual sessions), completers of the PM+ program will be randomized to receive a one-time booster session three months post-PM+, or to the control group, which will not receive the booster session. Both groups will be assessed at 3 months post-PM+ and 6 months post PM+ (the endline).
Masking Description: Because the intervention and control groups involve receiving or not receiving a booster session, neither participants nor providers can be blinded. Because the administration and data collection is being completed by the PI, who is also responsible for study administration, the PI cannot be blinded. Instead, randomization occurs after delivery of PM+ to avoid bias in PM+ delivery, and contact between the study administrator is limited to emailing questionnaires (with standardized language that does not differ between groups).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Booster Session Arm (Experimental): This group will receive a one-time PM+ booster session three months after finishing the PM+ program
  Interventions: Behavioral: Problem Management Plus booster session
- Control (No Intervention): This group will receive the full PM+ program but no booster session or meeting thereafter.

INTERVENTIONS:
Behavioral: Problem Management Plus booster session — A 60-minute session designed to refresh participants on the PM+ strategies (diaphragmatic breathing, problem management, behavioral activation, strengthening social support). Session consists of practicing strategies and developing plans for the future.
  Arms: Booster Session Arm

SUMMARY:
Therapists at the Grand Bahama Resilience Center (GBRC) will be trained to deliver Problem Management Plus (PM+), a WHO intervention. Then, those therapists will deliver PM+ (5 one-on-one skills-based sessions) to a total of 50 adult clients experiencing mild to moderate mental health difficulties (excluding anyone with cognitive difficulties or psychosis). Participants will complete (de-identified) self-report survey assessments before PM+, after PM+, 3 months later, and 6 months later. After receiving 5 sessions of PM+, participants will be randomized to either receive a one-time booster session of PM+ (to be co-created by the PI and the GBRC providers) three months later or to a control group which will receive a phone call reminding them that they will receive their third assessment soon.

DETAILED DESCRIPTION:
This mixed-methods study will consist of three overlapping phases. First, GBRC counselors will be trained to deliver PM+ ("GBRC providers"). After some experience with PM+ delivery and practice, researchers from The New School for Social Research will collaborate with GBRC providers to develop a protocol for a one-time PM+ booster session. Third, after receiving PM+, study participants will then be randomized to-at approximately three months post-PM+ -either receive the PM+ booster session, or to receive a phone call reminder of the upcoming electronic survey (the control group).

Fidelity to the intervention and booster session protocols will be measured via self-report checklists to be submitted by the provider at the conclusion of each session. After screening and informed consent, participants will be assessed for all outcome measures prior to receiving PM+, approximately one week post-PM+, approximately three months post-PM+, and approximately six months post-PM+. Qualitative interviews with participants will be conducted approximately one week after receiving the booster session, or one week after completing the three-month follow-up for control group participants, and at the six-month follow-up. Qualitative interviews with providers will take place after delivering the PM+ booster session and at the conclusion of data collection. An IRB application outlining all portions of the study will be submitted to BRANY through The New School for Social Research in the fall of 2024. Data collection will not commence until IRB approval is secured.

Participants Randomization will occur at the individual level. Participants will be adults (18 years or older) who reside in Grand Bahama and are recruited from visitors to the Grand Bahama Resilience Center (GBRC) in Freeport, Grand Bahama. Though PM+ is a transdiagnostic intervention, and therefore not intended to target specific disorders or symptoms, it is designed to help individuals who are experiencing psychological distress. The WHO PM+ manual recommends assessing potential PM+ clients using a measure of functioning such as the WHO disability assessment (WHODAS 2.0) and a measure of emotional distress such as the General Health Questionnaire (GHQ-12) or combining the Patient Health Questionnaire (PHQ-9) and the General Anxiety Disorder-7 (GAD-7) scale (WHO, 2016). The manual suggests using a cut-off score of ≥17 for the WHODAS and ≥10 for the PHQ-9 for inclusion, but does not offer guidance for other measures. Several past studies have used a cutoff score of ≥3 for the GHQ and the ≥17 for the WHODAS as inclusion criteria. Others have used the Kessler Psychological Distress Scale as a measure of emotional distress. For this study, following experiences of PM+ implementation in New York City, the Patient Health Questionnaire-4 (PHQ-4) will be used to assess for emotional distress and the self-report version of the Global Assessment of Functioning (GAF) will be used as a measure of functioning. Participants will be eligible for the study if they score ≥3 on the PHQ-4 and ≤90 on the GAF. Exclusion criteria will follow guidelines from the WHO PM+ manual and will include acute suicidality operationalized as "high risk" on the Columbia Suicide Severity Rating Scale (C-SSRS), active psychosis, or any impairment that would prohibit one from being able to engage in the intervention (e.g. cognitive disorder, substance use disorders; WHO, 2016). Procedure PM+ Provider Training Six experienced counselors working at the GBRC will be recruited as PM+ providers. Since these providers currently deliver counseling to community members, they will be referred to as "providers" rather than the more common term "helper" which typically connotes a non-mental health professional or a lay provider. Providers will undergo a 12-hour remote PM+ training, with weekly supervision meetings that will include ongoing PM+ education, expert supervision, and peer support. If a therapist decides to join the study at a later date, another 12-hour remote PM+ training will be conducted by the PI. The intensive training will take place between August and September of 2024 and will cover the PM+ protocol and procedures detailed in the WHO PM+ manual and will include modules on conducting the PSYCHLOPS assessment and suicide screening. Common therapeutic factors will be briefly noted, however, due to the experience level of the providers, this and other introductory material relating to working with clients in distress will be condensed. Researchers have found that 12 hours of PM+ helper training is sufficient for master's level social work students, therefore the same length should suffice for this group of providers. Training will include education on PM+ session agendas, strategies and rationales, and provider self-care. Competency and fidelity will be assessed pre- and post-training using the Ensuring Quality in Psychological Support (EQUIP) tool, a competency evaluation tool designed by the WHO specifically for task-sharing interventions such as PM+. Since its launch in 2022, the EQUIP tool has been used to assess provider competency in 36 countries throughout the world.

Booster Session Development Following training and initial delivery of PM+ to at least two clients, around approximately November-December 2024, researchers from The New School for Social research will meet with GBRC providers to develop a curriculum for a one-time PM+ booster session. The booster session will include a review of PM+ strategies and administration of Psychological Outcomes Profile (PSYCHLOPS) interview. The protocol and additional components of the booster session will be developed together with the GBRC providers, who are members of the Bahamian community and have experience delivering mental healthcare with the target population. Principles of CBPR will be used to ensure equitable contribution to all aspects of the protocol development. A deliverable of a supplementary chapter to the WHO PM+ manual will be created with authorship shared by academic and community partners.

Pilot Trial GBRC providers will recruit interested potential participants from their current clients and from their counseling waitlist. Upon obtaining IRB approval, approximately around early November 2024, eligible participants who complete informed consent will be invited to complete a baseline assessment in the form of a self-report Qualtrics survey. GBRC therapists will recruit particpants and will obtain informed consent from participants. Participants will then be assigned to a GBRC provider to receive PM+. As this study will be investigating the feasibility and acceptability of a booster session for clients who received the full 5-session course of PM+, both treatment arms will receive individual PM+ after enrollment. All participants will be emailed a post-treatment survey approximately one week after receiving PM+ (6-8 weeks after baseline).

Upon completing the fifth session of PM+, participants will be randomly allocated to either the booster group (i.e. treatment group) or the control group using block randomization. Blocks of four will be used and a random number generator will be used generate the block assignments. This ensures that providers are blinded to treatment groups during initial PM+ delivery (since they will not yet have been assigned) and it ensures that participants who do not complete PM+ are not included in randomization since they will not be eligible to continue in the study. Participants will be blinded to their allocated group (i.e. treatment or control) until they complete their final (6-month-follow-up assessment) or in the case that they drop out of the study. Blinding is necessary to the study to avoid a placebo effect for those in the treatment group. If participants were aware of their study group they may be influenced to practice or engage more with the intervention than if they are blinded to their condition. Moreover, because both groups will be contacted by their provider three months following the intervention-the control group for a phone call reminder of the upcoming third assessment, and the intervention group to conduct the booster session-the risks of harm by blinding are extremely low. All participants will be made aware of their group allocation (if applicable) at the conclusion of their involvement in the study and no later than July 31, 2026.

Participants who are randomized to the control arm will terminate treatment after their fifth session of PM+, and will be notified that they should complete three more online assessments. They will be told that they will receive the first of the remaining assessments in approximately one week, and to expect a phone call reminding them of the second of the remaining assessments in approximately three months.

Participants who are randomized to the PM+ with booster arm will meet with their provider approximately three months (beginning around March 2025) after their final PM+ session (17-19 weeks after their first PM+ session) for a one-time booster session. To ensure proper recollection of the booster session, a portion of the qualitative interviews with participants will take place one to three weeks after receiving the booster session of PM+. All participants will receive follow-up assessments approximately 17-19 weeks after their baseline assessment (3-month follow-up) and approximately 28-30 weeks after their baseline assessment (6-month follow-up). All follow-up assessments are to be completed by April 2026.

Qualitative interviews with providers will be conducted by research colleagues. Effort will be made to ensure that these interviewers are versed in cultural humility and ideally familiar with the Bahamian community. Client interviews will be conducted by trusted members of the Grand Bahama community including advanced social work students who have familiarity with PM+ and other Bahamian therapists not involved in the proposed study. Interviews with participants will take place on a rolling basis approximately one to three weeks after completion of the study protocol. Final qualitative interviews with providers will be completed no later than February and March 2026.

The GBRC will provide PM+ (without booster session) to clients regardless of involvement with the study. Clients who wish to receive PM+ but do not wish to participate in the study will be able to access that care and will not be penalized in any way. Study participants will not be prioritized over non-participant PM+ clients. Non-participant PM+ clients will receive standard PM+ according to the WHO manual, without the booster session as the booster session has not been formally studied and is therefore not currently evidence-based. Accordingly, clients who do not consent to participate in the study will not receive that experimental part of the program.

ELIGIBILITY:
Inclusion Criteria:

* Adults of 18 years or above

  * English-speaking
  * A score of <91 on Global Assessment of Functioning
* Located in the Bahamas

Exclusion Criteria:

* ● Imminent suicide risk (assessed at screening using Columbia Suicide-Severity Rating Scale, see document titled " Screener updated 10-30- 24")

  * Severe mental disorder (e.g. psychotic disorders)
  * Severe cognitive impairment (e.g. severe intellectual disability or dementia)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Hospital Anxiety and Depression Scale | From enrollment, again at week5, again at week 18 and finally at week 30
  Hospital Anxiety and Depression Scale (HADS) (Zigmond & Snaith, 1983) is a 14-item scale, which consists of two subscales of seven items each. One subscale measures symptoms of anxiety (HADS-A) and the other measures symptoms of depression (HADS-D). Responses are reported a four-point Likert scale, from 0-3, which pertain to different levels of symptom severity, depending on the question. Responses are summed to produce a total score, where higher scores indicate greater levels of anxiety and depression. Subscale scores may also be totaled to separate depression and anxiety symptoms. This scale has been used widely throughout the world and across many cultures, including in the US and in South America (Herrmann, 1997).

SECONDARY OUTCOMES:
PHQ-9 | At enrollment, again at week 5, again at week 18, and finally at week 30
  Patient Health Questionnaire (PHQ-9) (Kroenke et al., 1999) is a nine-item tool which measures depression severity. Responses are reported on a four-point Likert scale (from 0-3 with 0 indicating "not at all" and 3 indicating "extremely so"). Scoring is done by taking the sum of all nine items to produce a final score. Depression scores range from minimal (0-4), mild (5-9), moderate (10-18), moderately severe (19-26), to severe (≥27). While the PHQ-9 was designed as a diagnostic tool (Keoenke et al., 1999), it is frequently used to assess depression outcomes in studies of task-sharing interventions including PM+ (e.g., Rahman et al., 2016; Khan et al., 2019; Jordans et al., 2021; Nyongesa et al, 2022; Marchetti et al., 2024).
GAD-7 | At enrollment, again at week 5, again at week 18, and finally at week 30
  Generalized Anxiety Disorder Assessment (GAD-7) (Spitzer et al., 2006) is a seven-item tool designed to assess the severity of anxiety symptoms. Similar to the PHQ-9, responses are reported on a four-point Likert scale from 0-3 (with 0 indicating "not at all" and 3 indicating "nearly every day"). Responses are summed to produce a total final score. Scores indicate the severity of anxiety symptoms and range from minimal(0-4), mild (5-9), moderate (10-14), to severe (≥15). The GAD-7 is also commonly used to evaluate anxiety symptoms in studies of PM+ (Nyongesa et al., 2022; Luzano et al., 2023; Marchetti et al., 2024), despite being originally developed as a diagnostic tool (Spitzer et al., 2006)
PSYCHLOPS | At enrollment, at week 1, 2, 3, 4, and 18
  Psychological Outcomes Profile (PSYCHLOPS) (Ashworth et al., 2005) measures personally identified problems and stressors. The measure is administered as an interview and consists of four questions across three domains (problems, functioning, and wellbeing). Participants are asked to identify two problems, and one area of functioning in free-form text format. A six-point Likert scale (0-5) assesses how much the respondent has been affected by each. Respondents identify the problems and area of functioning at pre-intervention and are asked to assess each item during every session of PM+. In the proposed study, participants in the intervention arm will complete the PSYCHLOPS during the booster session as well. Scores are totalled and range from 0-20 with greater scores indicating greater distress related to personally identified problems.
PCL-5 | At enrollment, again at week 5, again at week 18, and finally at week 30
  PTSD Checklist for DSM-5 (PCL-5) (Weathers et al., 2013) is a 20-item checklist used to measure symptoms of PTSD based on the diagnostic criteria of the DSM-5. Each item is rated on a 5-point Likert scale (0-4, with 0 indicating "not at all" and 4 indicating "extremely"). Scores are summed and total scores range from 0-80 with higher scores indicating greater PTSD symptom severity. Following previous PM+ studies, the measure will be adapted to ask about symptoms in the past week rather than the past month to ensure sensitivity to detect changes at three- and six-month follow-ups.
WHODAS-2.0 | At enrollment, again at week 5, again at week 18, and finally at week 30
  WHO Disability Assessment Schedule (WHODAS-2.0) (Ütsün, 2010) is a 12-item tool used to assess functional impairment across six different domains of functioning (communication, hygiene and daily functioning, physical activity, interacting with others, domestic responsibilities, and participation in community activities). The proposed study will use the 12-item self-administered version of the WHODAS 2.0, wherein each item is rated on a 5-point Likert scale from 1-5 (with 1 indicating "none" and 5 indicating "extreme or cannot do"). Greater scores indicate more functional impairment.
GSES | At enrollment, again at week 5, again at week 18, and finally at week 30
  General Self Efficacy Scale (GSES) (Schwartzer & Jerusalem, 1995) is a 10-item scale, which measures one's overall sense of self-efficacy. Questions are scored on a 4-point Likert scale that ranges from "Not at all true" to "Exactly true," and then summed to produce a final score from 10 to 40. Higher scores indicate greater levels of perceived self-efficacy.
RTC | At enrollment, again at week 5, again at week 18, and finally at week 30
  Reducing Tension Checklist (RTC) (Jordans et al., 2021) is a 10-item tool used to measure the use of coping skills learned in PM+. Each of the four PM+ strategies (deep breathing for stress management, problem solving, behavioral activation, and strengthening social support) are assessed in items of the RTC. Scores are summed, resulting in a total score ranging between 0-40, with higher scores indicating greater use and practice of the intervention skills. The RTC was developed based on a coping checklist (Neacsiu et al., 2010). The measure was adapted to assess content specific to PM+ (Jordans et al., 2021).
PHDS | At enrollment
  Post-hurricane Distress Scale (PHDS) (Carl et al., 2019) is a 20-item survey that measures short- and long-term post-hurricane related stressors, which are known to affect mental health outcomes. The scale includes an initial occurrence item, in which respondents report whether they experienced the described item. Then, if endorsed, each item has a corresponding distress scale, in which respondents choose from a 5-item Likert scale from 1-5 (with 1 indicating "not at all bothered" and 5 indicating "extremely bothered"). Scores are totaled and range from 0-100 with a recommended cut-off score of 41 where scores greater than or equal to 41 indicate high risk for developing common mental health disorders including depression, anxiety, and PTSD.

CONTACTS AND LOCATIONS:
Overall Officials: Adam Brown D Brown, PhD, Study Chair — The New School
Locations (1):
- Grand Bahama Resilience Center, Freeport, Grand Bahama, The Bahamas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rahman A, Hamdani SU, Awan NR, Bryant RA, Dawson KS, Khan MF, Azeemi MM, Akhtar P, Nazir H, Chiumento A, Sijbrandij M, Wang D, Farooq S, van Ommeren M. Effect of a Multicomponent Behavioral Intervention in Adults Impaired by Psychological Distress in a Conflict-Affected Area of Pakistan: A Randomized Clinical Trial. JAMA. 2016 Dec 27;316(24):2609-2617. doi: 10.1001/jama.2016.17165. PMID 27837602
- [Background] Dawson KS, Bryant RA, Harper M, Kuowei Tay A, Rahman A, Schafer A, van Ommeren M. Problem Management Plus (PM+): a WHO transdiagnostic psychological intervention for common mental health problems. World Psychiatry. 2015 Oct;14(3):354-7. doi: 10.1002/wps.20255. No abstract available. PMID 26407793
- [Background] Bryant RA, Schafer A, Dawson KS, Anjuri D, Mulili C, Ndogoni L, Koyiet P, Sijbrandij M, Ulate J, Harper Shehadeh M, Hadzi-Pavlovic D, van Ommeren M. Effectiveness of a brief behavioural intervention on psychological distress among women with a history of gender-based violence in urban Kenya: A randomised clinical trial. PLoS Med. 2017 Aug 15;14(8):e1002371. doi: 10.1371/journal.pmed.1002371. eCollection 2017 Aug. PMID 28809935
- See also: Link to PM+ Manual — https://www.who.int/publications/i/item/WHO-MSD-MER-18.5